CLINICAL TRIAL: NCT02352142
Title: Randomized Control Trial of Family Nurture Intervention in the Children's Hospital of New Jersey Neonatal Intensive Care Unit
Brief Title: Family Nurture Intervention in the CHoNJ NICU
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient enrollment numbers
Sponsor: Columbia University (Other)
Collaborators: Newark Beth Israel Medical Center (Other)
Responsible Party: Principal Investigator, Martha G. Welch, MD, Assistant Professor, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AAAN6850
Record Dates: First submitted 2015-01-16; First posted 2015-02-02 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2016-07

CONDITIONS: Premature Birth
Keywords: Separation stress; Family Nurture; Maternal Confidence; Maternal Competence; Calming Cycle; Kangaroo Care; Infant Neurodevelopment; Infant Psychological Development; Post-partum depression; Mother-infant Co-regulation
MeSH Terms: conditions — Premature Birth; Depression, Postpartum

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard Care (No Intervention): Mothers are given infant care instruction as part of standard care
- Facilitated infant care (Experimental): Family Nurture Intervention
  Interventions: Behavioral: Facilitated Infant Care
- Full Term EEG (Other): Small group of healthy, Full-Term infants will receive two sleep EEGs (one in unit, and one 4 weeks post discharge) for healthy control comparison to preterm infants
  Interventions: Other: Full Term EEG

INTERVENTIONS:
Other: Full Term EEG — Full-term infants assigned to this arm of the study will receive one sleep EEG (one hour in duration). These EEGs will be used as healthy control comparisons to those of premature infants at 40 weeks.
  Arms: Full Term EEG
Behavioral: Facilitated Infant Care — Family Nurture Intervention is facilitated by specially trained Nurture Specialists. The intervention involves calming interactions between mother and infant in the isolette via odor exchange, firm sustained touch and vocal soothing, through calming interactions during holding and feeding via the Calming Cycle and through family sessions designed to engage the help and support of family members for the mother.
  Other Names: Family Nurture Intervention
  Arms: Facilitated infant care

SUMMARY:
The purpose of this proposal is to conduct a replication study of Family Nurture Intervention (FNI) at CHoNJ. FNI facilitates mother-infant interactions that are vital to early development. These include early and repeated mother/infant calming interactions during the NICU stay, such as interactive touch with vocal soothing, sustained reciprocal olfactory exposure and family practice in comforting, and systematically implemented skin to skin holding. This has already been studied at CHONY. Findings reveal that infants who receive FNI have significant increases in EEG power, a measure of brain activity, near to term age, when compared with those who receive Standard Care.

There will be two groups; STANDARD CARE (SC) and INTERVENTION (FNI). In addition, 10 pilot subjects will be enrolled to train the staff involved in the procedures used in this Randomized Control Trial (RCT). The pilot patients will be enrolled identical to study patients and will be encouraged to participate fully. They will not be included in the analysis of the RCT.

The STANDARD CARE group will receive current standard of care in NICU. The INTERVENTION group, in addition to the standard care, will receive the FNI intervention, which will be facilitated by our Nurture Specialists. In addition to the SC and FNI groups, there will be a third non-randomized group of infants born at term age who will receive standard care for newborns at CHoNJ. Assessments in the NICU will include physiological measures (ECG EEG), measures of maternal sensitivity through recorded mother-infant interactions and a variety of specimen collections (saliva, blood, and breast milk samples). The investigators will be conducting two follow up studies, at 4 months corrected age and at 12 months corrected age. The investigators will test the immediate and long-term effects of this approach to the development of preterm infants.

The investigators hypothesize that this intervention will alter a wide range of indices of physiological regulatory capacities, and increase brain activity as measured by EEG (power and coherence) such that a brain activation pattern in the intervention group will be more similar to that of full term infants as opposed to the standard care group. Longer term indices of mother psychological and infant neurobehavioral outcomes will also be improved when assessed during the first few months of life.

DETAILED DESCRIPTION:
The purpose of this study is to compare the value of the current approach of encouraging contact between mothers and their babies (Standard Care) in the NICU with a more wide ranging enhanced approach (Family Nurture Intervention). This approach is based on enhancing aspects of maternal nurturing including mother-infant reciprocal calming, which are vital to early development. A specific goal is to improve the mother's view of her baby, reduce negative emotions about having delivered a baby prematurely, and help her gain confidence in her caretaking abilities. Since preterm babies are often easily upset, this study will facilitate mothers in comforting and calming their babies. An earlier study at Morgan Stanley Children's Hospital of New York (CHONY) has shown positive outcomes in the enhanced treatment group in a variety of areas, including EEG brain activity at term age. Assessments in the NICU and in secondary follow-up measures at 4, and 12 months of age will test the immediate and long-term effects of this new enhanced approach to the nurture of prematurely born infants. We will undertake a replication study on patients in the NICU at CHoNJ to confirm and further elucidate the positive effects of enhanced nurturing.

We hypothesize that enhanced nurturing will alter a wide range of physiologic regulatory capacities, reduce morbidity, decrease Length of Stay (LOS) and increase brain activity as measured by EEG (power and coherence). In addition this approach may influence a brain activation pattern (particularly in the area of the anterior cerebral cortex responsible for executive decision-making) in the intervention group that is more similar to that of a full term infant. Longer term measures of mother's psychological and infant's neurobehavioral outcomes will also be improved when assessed during the first few months of life.

This study aims to replicate and build on an existing study at Morgan Stanley Children's Hospital of New York (CHONY) that compares the current protocol for encouraging mother/infant interactions (standard care) with a multifaceted intervention to enhance mother and infant bonding (Family Nurture Intervention - FNI). The FNI was piloted and studied in a cohort of 150 mother-infant pairs at CHONY beginning in 2009. While the study is ongoing, significant differences in brain activity of these preterm infants was found at term as measured by EEG power in the intervention premature infants as compared to the standard care group, with no increased risk of morbidity or mortality in the intervention group. The study demonstrated that the approach may influence a brain activation pattern (particularly in the area of the anterior cerebral cortex responsible for executive decision-making) in the intervention group that is more similar to that of a full term infant (38-42 weeks gestation).

This and other research warrants the investigation of better intervention strategies that can reduce morbidity and ameliorate adverse outcomes in these infants.

The purpose of this current study is to determine whether the findings from CHONY are replicable, the efficacy of the FNI protocol in improving developmental outcomes in preterm births in a different cohort (at CHoNJ) and to compare the outcomes of patients in two different hospital environments.

The study will again compare the current standard of care in the NICU, which includes periodic skin-to-skin holding, to a Family Nurture Intervention (FNI) which adds other interventions: interactive touch with vocal soothing, sustained reciprocal olfactory exposure, and family modeling and practice in comforting as well as a more systematic implementation of skin-to-skin holding. The behavioral, neurobiological and clinical insights gained from this project may eventually lead to better prevention of developmental disorders, reduced morbidity and more effective clinical intervention strategies both in the neonatal intensive care unit (NICU) and after discharge. We hypothesize that the treated babies will show better results in the primary outcome measure in the short term and secondary long term as compared to infants undergoing standard care.

ELIGIBILITY:
Inclusion Criteria:

* Infant is between 26/0 and 32/6 weeks gestational age upon admission for the INTERVENTION / STANDARD care group OR 38-42 weeks for the FULL TERM group
* Infant's weight is appropriate for gestational age (AGA)
* Infant is a singleton
* Mother is 18 years of age or older
* Mother has at least one supporting person in the home (e.g. significant other, mother, father, sibling, aunt, grandmother, step-parent) (not applicable for FULL TERM group)

Exclusion Criteria:

* Infant's attending does not recommend enrollment in study
* The infant has severe congenital anomalies, including chromosomal anomalies or an Intraventricular Hemorrhage (IVH) Grades 3 and 4
* Mother has known history of substance abuse, severe psychiatric illness or psychosis
* Status of enrolled subject changes and subject no longer falls in inclusion criteria
* Mother and/or infant has a medical condition that precludes intervention components
* Mother and/or infant has a contagion that endangers other participants in the study
* Mother-Infant dyad receives less than one week of intervention (not applicable to the FULL TERM group)

Ages: 26 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2015-01; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
EEG measures of power and coherence | 34 weeks gestational age through term age
  Two one-hour sleep EEGs will take place. One at 34-36 weeks Gestational Age, and one at term age

SECONDARY OUTCOMES:
Maternal measures of anxiety, depression and care-giving | Up to 12 months of age
  Measures of maternal depression and anxiety and maternal care-giving will be compared between standard care and intervention groups using analyses of variance. The measures will also be compared within groups, using repeated measures ANOVA.
Measure of mother time spent with infant in unit and in skin to skin | Duration of infant stay in unit (roughly 35 days)
  Measures of parental visiting hours and occurrence of skin to skin will be compared within groups. We will use parent and nurture specialist report to measure parental visiting hours and occurrence of skin to skin.
Neurobehavioral Assessments of Infants- Bayley Scales of Infant and Toddler Development, Bayley III | Up to 12 month corrected age
  At 4 and 12 months corrected age, infants are administered the Bayley Scales of Infant and Toddler Development, Bayley III consisting of four subscales: Cognitive, Language (receptive/expressive), Motor (fine/gross) and Social-Emotional. These filmed assessments, made by research staff 'blind' to infant group assignment, provide information about the neurobehavioral status of the child and whether there are significant delays in key domains of motor, language, and cognitive development.
Physiological Assessments- salivary cortisol | Up to 24 months corrected age
  As a component of the mother-infant interaction assessments conducted at 4 and 12 months corrected age, salivary cortisol levels are measured at four times during each session. These measures provide physiological indices of how the infants respond to a social interaction stressor.
Physiological Assessments- breast milk | The duration of the infant stay in unit, or an average of 5 weeks
  Breast milk collections will be analyzed in order to measure levels of pro-inflammatory cytokines, oxytocin and other peptides.
Physiological Assessments- infant stool collection | The duration of the infant stay in unit, or an average of 5 weeks
  Infant stool collections will be made in order to measure levels of inflammation-related cytokines and other peptides.
Physiological Assessments- infant blood samples | The duration of the infant stay in unit, or an average of 5 weeks
  Infant blood samples will be collected by piggy-backing off of standard care heel-sticks by hospital staff. These samples will be analyzed for presence of oxytocin and other applicable peptides
Mother-Infant Interactions Assessments: Evaluating the qualities of the mother's interaction with her infant during diaper change | Up to 4 months corrected age
  Videos of infant's diaper change are obtained and coded by research team members unfamiliar with the dyads' group assignment at 4 months corrected age. The mother is instructed to undress her infant, remove the diaper, wipe clean, and re-dress her infant. These familiar caregiving procedures represent a mild, ecologically valid stressor. Maternal behavior is coded, using a 9-point Likert scale for: (a) Acceptance vs. Rejection; (b) Soothing capability; (c) Consideration vs. Intrusiveness; (d) Quality of Physical Contact; and (e) Quality of Vocal Contact.
Mother-Infant Interaction Assessments: Mother-infant face-to-face communicative competence, sensitivity of maternal caregiving and mother and infant physiological capacity to cope with a stressor | Up to 12 months corrected age
  A split-screen filming session is conducted following protocols and analyzed by team members 'blind' to the dyads' group assignments at 4, 12, and 24 months corrected age. The videotapes consist of: (1) mother-infant play; (2) stranger-infant play (3) diaper change; (4) the Still Face protocol in which mothers assume an expressionless face for two minutes. Primary measures are: infant gaze aversion, mother-infant gaze coordination, infant distress, maternal interaction style (affectionate vs. intrusive), and responses of mothers and infants to gaze aversion. Additionally, research staff blind to group assignment will assess the quality of the mother-infant interaction with the Biphasic Emotional Connection Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Martha G Welch, MD, Principal Investigator — Columbia University Medical Center, Presbyterian Hospital
Locations (2):
- United States (2):
  - Children's Hospital of New Jersey, Newark, New Jersey
  - Columbia University Data Coordinating Center, New York, New York

REFERENCES:
- [Background] Ravn IH, Smith L, Lindemann R, Smeby NA, Kyno NM, Bunch EH, Sandvik L. Effect of early intervention on social interaction between mothers and preterm infants at 12 months of age: a randomized controlled trial. Infant Behav Dev. 2011 Apr;34(2):215-25. doi: 10.1016/j.infbeh.2010.11.004. Epub 2011 Mar 2. PMID 21371754
- [Background] Muller-Nix C, Forcada-Guex M, Pierrehumbert B, Jaunin L, Borghini A, Ansermet F. Prematurity, maternal stress and mother-child interactions. Early Hum Dev. 2004 Sep;79(2):145-58. doi: 10.1016/j.earlhumdev.2004.05.002. PMID 15324994
- [Background] Meijssen D, Wolf MJ, van Bakel H, Koldewijn K, Kok J, van Baar A. Maternal attachment representations after very preterm birth and the effect of early intervention. Infant Behav Dev. 2011 Feb;34(1):72-80. doi: 10.1016/j.infbeh.2010.09.009. Epub 2010 Nov 9. PMID 21067812
- [Background] Meijssen D, Wolf MJ, Koldewijn K, Houtzager BA, van Wassenaer A, Tronick E, Kok J, van Baar A. The effect of the Infant Behavioral Assessment and Intervention Program on mother-infant interaction after very preterm birth. J Child Psychol Psychiatry. 2010 Nov;51(11):1287-95. doi: 10.1111/j.1469-7610.2010.02237.x. PMID 20345840
- [Background] Shah PE, Clements M, Poehlmann J. Maternal resolution of grief after preterm birth: implications for infant attachment security. Pediatrics. 2011 Feb;127(2):284-92. doi: 10.1542/peds.2010-1080. Epub 2011 Jan 17. PMID 21242223
- [Background] Coppola G, Cassibba R, Costantini A. What can make the difference? Premature birth and maternal sensitivity at 3 months of age: the role of attachment organization, traumatic reaction and baby's medical risk. Infant Behav Dev. 2007 Dec;30(4):679-84. doi: 10.1016/j.infbeh.2007.03.004. Epub 2007 Apr 20. PMID 17449102
- [Background] DeBoer RW, Karemaker JM, Strackee J. Comparing spectra of a series of point events particularly for heart rate variability data. IEEE Trans Biomed Eng. 1984 Apr;31(4):384-7. doi: 10.1109/TBME.1984.325351. No abstract available. PMID 6745974
- [Background] Hofer MA. Early social relationships: a psychobiologist's view. Child Dev. 1987 Jun;58(3):633-47. PMID 3608643
- [Background] Als H, Lawhon G, Duffy FH, McAnulty GB, Gibes-Grossman R, Blickman JG. Individualized developmental care for the very low-birth-weight preterm infant. Medical and neurofunctional effects. JAMA. 1994 Sep 21;272(11):853-8. PMID 8078162